CLINICAL TRIAL: NCT05562427
Title: Using Multimodal Real-Time Assessment to Phenotype Dietary Non-Adherence
Brief Title: Program for Fully Understanding Eating and Lifestyle Change (FUEL)
Acronym: FUEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stephanie Goldstein, Research Scientist, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DK132210 (NIH); R01DK132210 (NIH)
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Obesity
Keywords: Diet; Digital health; Ecological momentary assessment; Behavioral phenotyping; Wearable sensors; Geolocation; Smartphone; Passive sensing; Eating behavior
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1 (Other): Gold-standard online behavioral weight loss treatment
  Interventions: Behavioral: Gold-Standard Online Behavioral Obesity Treatment

INTERVENTIONS:
Behavioral: Gold-Standard Online Behavioral Obesity Treatment — Rx Weight Loss (RxWL) is an online BOT that consists of: (a) tailored weight loss, calorie, and physical activity goals. (b) 12 weekly 10-15 minute multimedia lessons for training in behavioral weight loss skills followed by 9 monthly lessons for continued weight loss. Lessons incorporate video, animation, audio, quizzes, and exercises for goal setting, planning, and problem-solving. Example topics include restaurant eating, changing the home environment, and obtaining social support. (c) Online tools for self-monitoring weight, diet, and physical activity that interface with popular tracking apps; and (c) Weekly, and eventually monthly, automated feedback on progress to date (delivered as text appearing on the platform). If goals are not met participants receive strategies to improve weight loss, along with encouragement. To ensure engagement, email reminders are sent to participants who have not visited the platform on a given week.
  Other Names: Rx Weight Loss (RxWL)

SUMMARY:
This project seeks to better understand dietary lapses (instances of nonadherence to dietary goals), a major cause of poor outcomes during behavioral obesity treatment (BOT). Investigators propose to conduct multimodal real-time assessment of behavioral, psychosocial, and contextual characteristics to uncover lapse phenotypes (i.e., meaningful clusters of lapse behaviors, such as lapsing via overeating vs. lapsing via eating an off-plan food). Using wearable sensors and a smartphone-based assessment platform, this research will identify latent characteristics underlying different phenotypes of dietary lapses reported by individuals who are participating in an online BOT. This study will also evaluate how these emerging lapse phenotypes vary over time, between individuals, and within individuals. Such information will ultimately help the field understand how best to reduce lapses in future treatments (e.g., how much to personalize future interventions for lapse vs. generalizability of lapse phenotypes across individuals). Therefore, this study has three goals. First, investigators aim to establish lapse phenotypes by identifying clusters of behavioral, psychosocial, contextual and individual-level factors (e.g., sex, race) that differentiate lapse behaviors during weight loss and maintenance. Second, the investigators aim to test the association of lapse phenotypes with energy intake and weight change during weight loss and maintenance to determine which lapse phenotypes have the greatest impact on BOT outcomes (e.g. personal, environmental, and behavioral factors). Lastly, investigators aim to evaluate individual variability in the occurrence of lapse phenotypes during weight loss and maintenance to determine the generalizability of lapse phenotypes across individuals.

Participants will be recruited through various methods including advertisements in local media, targeted online advertising, advertisements in medical and minority communities, and direct mailers. All participants will receive a well-established online BOT program for 12 months, with a 6-month maintenance period, for a total study participation of 18 months. In conjunction, they will complete 14-day monitoring periods (at baseline, 3 months, 6 months, 12 months, and 18 months) consisting of: 1) repeated daily smartphone surveys to assess personal, environmental, and behavioral factors, including automatic capture of geographic location; 2) wearing two wrist-based sensor devices to passively capture physical activity, sleep, and eating behaviors; and 3) completing telephone-based 24-hour dietary recalls to assess overall energy intake. Weight will be measured at all visits to the research center.

DETAILED DESCRIPTION:
The purpose of this 5-year study is to conduct multimodal real-time assessment of behavioral, psychosocial, and contextual characteristics to uncover lapse phenotypes. The data from this project will ultimately inform future personalized interventions to promote dietary adherence by providing critical data on which lapses to target and how to best target them. Participants (N=150) will receive 12 months of online behavioral obesity treatment followed by a 6-month maintenance period (18 months of study participation total). The primary aim is to establish lapse phenotypes by identifying clusters of factors that differentiate lapse behavior. The secondary aim is to evaluate associations of emerging lapse phenotypes with clinical outcomes (e.g., energy intake and weight loss). The investigators will also explore the variability in lapse phenotypes based on data collected from the primary outcome.

Participants will be recruited on a rolling basis until the target (N=150) is reached. Participants will be recruited via advertisements in local media (e.g. newspapers, radio) and online advertising (e.g., Google AdWords, social media), flyers and advertisements posted in waiting rooms and exam rooms in primary care offices, informational materials made available as part of the health and wellness program for employees in the Lifespan hospital network, and direct mailings.

Interested individuals will be initially screened for eligibility via REDCap (a Lifespan secure website) or via telephone. If a participant appears to be eligible based on their responses to the screening questions, they will receive a follow-up call from the research team to confirm eligibility, describe the study in more detail, and schedule an orientation meeting. If they are not eligible, they will receive a message indicating that they are not eligible for the study and directed to contact the research team if they wish to receive referrals for other weight loss programs. Those who are eligible will be invited to an orientation via the online video chat forum Zoom, where the study will be described, and informed consent obtained. Only after the consent form is signed will any further study procedures be completed. If consent is not given, participant contact information will be immediately removed from the system. After consent is obtained, participants will complete baseline questionnaires via REDCap. Paper surveys will be made available for participants who prefer this option. If a participant elects to use a paper questionnaire, the questionnaire will be sent to the participant's home address. Participants will then complete a 1-week behavioral run-in in which they complete smartphone-based surveys and wear the sensors. This data is for testing only and will not be used in the analysis of primary outcomes. Participants must complete >70% of EMA surveys and wear both devices >10 hrs/day to move forward with the remainder of study procedures. Following consent and successful completion of baseline procedures, participants will attend an in-person "kick-off" session to assist them in using the online BOT program. Participants will be given access to an online BOT (described further in the Intervention section) for 12 months, with an additional 6 months of no treatment follow-up (intended to serve as a weight maintenance period).

During this 18-month study period, participants will complete 5 total assessments at baseline, 3, 6, 12, and 18 months. Each assessment consists of a 14-day monitoring period. There will be 2 visits with trained research staff at the beginning and end of the 14-day monitoring. At the first visit, participants will: have their height/weight measured, receive study equipment (e.g., wearable wrist devices), and undergo training in using study equipment. Participants will be instructed to wear the sensor devices, complete repeated smartphone surveys for 14 days, and complete three non-consecutive telephone-based 24-hour dietary recalls with staff. At the end of 14 days, participants will return for their second visit in which they will: have their weight measured, return study equipment, and receive payment. The research staff do not need to be blinded for study visits because all participants are assigned to the same intervention. Participants will be asked to complete the same assessment procedures at baseline (first two weeks of the online BOT), 3, 6, 12, and 18 months (last two weeks of no- treatment weight maintenance period).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70
* Body mass index (BMI) between 25 and 50 kg/m-squared

Exclusion Criteria:

* Has health problems for which weight loss or physical activity is contraindicated
* Currently pregnant or breastfeeding
* Currently or recently (< 6 months) enrolled in a commercial weight loss program
* Weight loss of ≥ 5% of initial body weight in the last 6 months
* Currently taking weight loss medication,
* Has history of surgical procedure for weight loss,
* Has history of a clinically diagnosed eating disorder excluding Binge Eating Disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in dietary lapses | Baseline, 3 months, 6 months, 12 months, and 18 months
  Smartphone-based ecological momentary assessment (EMA) surveys will be used to assess dietary lapses, defined as exceeding a pre-planned calorie target for a given meal or snack. Participants will be asked to report if they experienced a "dietary lapse" since the last EMA survey. Participants can also initiate a report of a dietary lapse at any time. Participants will also record the time that the lapse occurred. Participants will be asked "how would you describe the lapse?" and can select all that apply from: 'I ate a larger portion', 'I ate when I hadn't intended', 'I ate a type of food I wanted to avoid', 'I planned to lapse', 'I did not know the calories in the food.'

SECONDARY OUTCOMES:
Change in weight | Baseline, 3 months, 6 months,12 months, and 18 months
  Weight will be measured by trained research staff at the research center to the nearest 0.1 kg using a calibrated digital scale. Measurements will be made in light indoor clothing without shoes.
Change in energy intake | Baseline, 3 months, 6 months, 12 months, and 18 months
  Participants will complete 3 non-consecutive telephone-based 24-hour dietary recalls. Recalled intake will be collected over 2 weekdays and 1 weekend day. The Nutrition Data System for Research (NDSR), a software application developed at the University of Minnesota Nutrition Nutrition Coordinating Center (NCC), will facilitate collection of recalls in a standardized fashion. Dietary intake interviews will be governed by a multiple-pass interview approach during which participants receive 5 opportunities to recall food intake. Recalled intake and independently observed intake are highly correlated, indicating the 24-hour dietary recall is highly valid and considered the goal-standard of dietary assessment. NDSR will generate daily estimates of usual energy intake using the NCC Food and Nutrient Database.

OTHER OUTCOMES:
Height | Baseline, 3 months, 6 months, 12 months, and 18 months
  Height will be measured by trained research staff at the research center in millimeters using a wall-mounted stadiometer. Measurements will be made without shoes.
Change in affect levels | Baseline, 3 months, 6 months,12 months, and 18 months
  Affect will be assessed via an adapted Positive and Negative Affect Schedule (PANAS) that was validated for use in EMA. Participants rate items on a scale from 1 (not at all) to 100 (very much), with 100 meaning they are experiencing the emotion to a more intense degree.
Change in energy levels | Baseline, 3 months, 6 months,12 months, and 18 months
  Energy levels will be assessed via items from the adapted PANAS, as above, that was validated for use in EMA. Participants rate items on a scale from 1 (not at all) to 100 (very much), with 100 meaning they are having that particular experience to a more intense degree.
Change in stress levels | Baseline, 3 months, 6 months,12 months, and 18 months
  Stress will be assessed during each EMA survey with 3 items of the Perceived Stress Scale, adapted for EMA by prior research. Participants rate items on a scale from 1 (not at all) to 100 (very much), with 100 indicating a greater degree of stress.
Change in motivation levels | Baseline, 3 months, 6 months,12 months, and 18 months
  Consistent with prior studies using EMA to evaluate the role of motivation in appetitive behaviors, motivation will be assessed by 1 item at each EMA survey: "How committed are you to your weight control goals for the rest of the day?", rated on a scale from 1 (not at all) to 100 (extremely).
Change in self-efficacy | Baseline, 3 months, 6 months,12 months, and 18 months
  Consistent with prior studies using EMA to evaluate the role of self-efficacy in appetitive behaviors, self-efficacy will be assessed by 1 item at each EMA survey: "How confident are you in your ability to succeed in your weight control goals?", rated on a scale from 1 (not at all) to 100 (extremely).
Change in distorted thinking patterns | Baseline, 3 months, 6 months,12 months, and 18 months
  After reporting an eating episode, participants will be asked the following 2 questions via EMA, adapted from the Dichotomous Thinking in Eating Disorders Scale and used in prior EMA research on lapse behaviors: "I feel like giving up my diet plan" and "I feel I have failed my diet plan", both rated on a scale of 1 (Strongly Disagree) to 100 (Strongly Agree).
Change in self-compassion | Baseline, 3 months, 6 months,12 months, and 18 months
  After reporting an eating episode, participants will be asked the following 3 items via EMA, taken from the Self-Compassion Scale- Short Form, adapted for EMA in prior research: 'I have been obsessing and fixating over breaking my diet', 'I have been understanding about breaking my diet', and 'I have been judgmental about breaking my diet', all rated on a scale from 1 (Strongly Disagree) to 100 (Strongly Agree).
Change in executive functioning | Baseline, 3 months, 6 months,12 months, and 18 months
  Executive function will be assessed at each survey via 4 items from the Quality of Life in Neurological Disorder short form item bank, each rated on a scale from 1-100 with higher scores indicating more impaired executive function.
Change in homeostatic hunger | Baseline, 3 months, 6 months,12 months, and 18 months
  Homeostatic hunger will be assessed at each EMA survey by asking "Please rate the extent to which you feel physically hungry right now", rated from 1 (not at all) to 100 (extremely).
Change in hedonic hunger | Baseline, 3 months, 6 months,12 months, and 18 months
  Hedonic hunger will be measured at each EMA survey using items from the Power of Food Scale, adapted for EMA. Participants will rate items on a scale of 1-100, with 100 indicating a higher degree of hedonic hunger.
Change in satiety | Baseline, 3 months, 6 months,12 months, and 18 months
  Satiety will be measured at each EMA survey via 4 items concerning appetite (I am full, I am satisfied with the amount of food I have eaten, I have a desire to eat, I think I could eat right now), rated on a scale from 1 (not at all) to 100 (extremely).
Change in food cravings | Baseline, 3 months, 6 months,12 months, and 18 months
  Food cravings will be assessed via 1 item at each EMA survey, "How strong is your craving to eat a specific food right now?", rated from 1 (low intensity) to 5 (high intensity). This measure is consistent with our prior work as well other previously published EMA studies of cravings.
Change in dietary composition | Baseline, 3 months, 6 months,12 months, and 18 months
  After reporting an eating episode, participants will be asked via EMA to indicate the types of foods consumed from a checklist (e.g., fruits and vegetables, starchy foods, fish, meat, poultry, cheese, sweets or chocolates, crisps/savory snacks) based on the Dietary Targets Monitor.
Change in alcohol intake | Baseline, 3 months, 6 months,12 months, and 18 months
  Consistent with prior EMA studies of alcohol intake, participants will be asked at each EMA survey if they consumed alcohol since the prior EMA survey and, if yes, they will be asked how many drinks were consumed.
Change in social support | Baseline, 3 months, 6 months,12 months, and 18 months
  Consistent with prior EMA work investigating the associations between social context and eating behavior more generally, participants will be asked the following when reporting a lapse via EMA: "When you lapsed, were there people eating?" (response options: 'no', 'yes, in my group', and 'yes, in view'), "Did others approve of your eating?" and "Did others encourage you to eat?" (response is a 0-100 scale agreement rating for both).
Change in television watching habits | Baseline, 3 months, 6 months,12 months, and 18 months
  Consistent with our prior studies, and the work of others, television use will be assessed at each EMA survey if the participant has watched television (or subscription online streaming equivalent) since the last survey.
Change in immediate food availability | Baseline, 3 months, 6 months,12 months, and 18 months
  The presence of tempting high-calorie foods and healthy foods (defined as the food being visible and accessible to eat) will be assessed at each EMA survey as in previous studies. If participants respond 'yes' to any food being available, they will be given a follow-up question, "Did any of the following make it easier for you to eat or drink", with a checklist that includes items related to food expense and social factors.
Change in adherence to Behavioral Obesity Treatment | Baseline, 3 months, 6 months,12 months, and 18 months
  The online behavioral obesity treatment will automatically record which lessons have been viewed by the participant each week and the number of days in which participants self-monitored diet, physical activity, and weight each week.
Demographic Information | Baseline
  The following will be assessed via questionnaire: age, sex, race, ethnicity, nativity, martial/relationship status, occupational status, level of education, and household income.
Change in basal metabolic rate | Baseline, 3 months, 6 months, 12 months, and 18 months
  The Harris-Benedict equation, which uses height, weight, age, and sex to estimate basal metabolic rate, will be used. Previous studies have shown that the Harris-Benedict equation yields high agreement with a handheld indirect calorimeter.
Neighborhood Socioeconomic Position | Baseline
  The participant's home address will be used to determine neighborhood socioeconomic position. Census tracts will be used as the participant's neighborhood unit. Census tracts are a useful proxy of neighborhood, and are widely applied in the health epidemiology literature. Census tracts will be used to extract median household income and proportion of the population whose ratio of income to poverty level is 100% below the federal poverty line.
Change in objective eating behavior | Baseline, 3 months, 6 months,12 months, and 18 months
  Participants will wear the ActiGraph GT9X Link on their dominant wrist (of the hand they typically eat with) daily, during waking hours, for the 14-day assessment period. This ActiGraph uses an inertial measurement unit (IMU) to detect the wrist-roll motion of food being brought to the mouth. In prior work, IMU data have been used to infer when someone is eating (in the field - during daily life, not in lab) with 89% accuracy, as well as accurately detecting 86% of bites taken during a detected eating event.
Change in objective physical activity | Baseline, 3 months, 6 months,12 months, and 18 months
  Participants will wear the ActiGraph xGT3X-BT on the non-dominant wrist to measure physical activity. Participants will wear this device 24/hours per day during each assessment period. The ActiGraph uses a 3-axis accelerometer to accurately and reliably measure physical activity among adults during daily life. Validated cutpoints will be used to categorize and timestamp bouts of physical activity for use in analysis. Consistent with prior work, vector magnitude counts per minute thresholds (shown to minimize mean differences of wrist vs. hip-based measurements) will be applied to estimate time spent at varying activity intensities: 2000-7500 counts = light and > 7500 counts = moderate-to-vigorous intensity activity. These data will be used to estimate physical activity just before and after a lapse, as well as total daily activity minutes.
Change in objective sedentary behavior | Baseline, 3 months, 6 months,12 months, and 18 months
  Validated cutpoints will be used to categorize and timestamp bouts of sedentary time from the ActiGraph GT3X (above) for use in analysis. Consistent with prior work, <2000 vector magnitude counts per minute thresholds (shown to minimize mean differences of wrist vs. hip-based measurements) will be considered as sedentary time. These data will be used to estimate sedentary behavior just before and after a lapse, as well as total daily sedentary minutes.
Change in objective sleep time | Baseline, 3 months, 6 months, 12 months, and 18 months
  The ActiGraph xGT3X-BT (worn on the non-dominant wrist as above) will be also used to measure sleep behaviors. The ActiGraph combines 3-axis accelerometer measurements and ambient light sensors to produce validated estimates of sleep behaviors. Cole-Kripke and Tudor-Locke algorithms will be used within ActiGraph software (ActiLife) to infer sleep periods.
Change in objective sleep efficiency | Baseline, 3 months, 6 months, 12 months, and 18 months
  The ActiGraph xGT3X-BT (worn on the non-dominant wrist as above) will be also used to measure sleep behaviors. The ActiGraph combines 3-axis accelerometer measurements and ambient light sensors to produce validated estimates of sleep behaviors. Cole-Kripke and Tudor-Locke algorithms will be used within ActiGraph software (ActiLife) to infer sleep efficiency (i.e., time spent asleep vs. time spent in bed).
Change in location | Baseline, 3 months, 6 months,12 months, and 18 months
  A smartphone based assessment used to facilitate EMA data collection, will also be used to collect near-continuous objective location data. The smartphone-based EMA platform will use smartphone global positioning system (GPS) receivers to capture geographic location (i.e., latitude and longitude coordinates). Previous research has demonstrated that smartphone GPS systems have a high degree of positional accuracy and are therefore appropriate for use in the proposed research. GPS coordinates will be analyzed with geographic information systems (GIS) software to interpolate participant location (particularly whether they are at home, work, restaurant, or other eating location).
Change in food accessibility | Baseline, 3 months, 6 months,12 months, and 18 months
  Smartphone-measured GPS coordinates, collected as described directly above ("Geolocation"), can also be used to infer food accessibility. GIS software will be used to develop an extensive database of addresses of food sources in the Rhode Island/Massachusetts area (location of the primary data collection site). Consistent with prior epidemiological research on food environment and availability, GPS coordinates collected via smartphone will be analyzed and combined with the established database of known food sources to calculate the following for each measured location point: least-cost driving proximity to food sources and density of food sources within a 0.5 mile radius.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstein SP, Mwenda KM, Hoover AW, Shenkle O, Jones RN, Thomas JG. The Fully Understanding Eating and Lifestyle Behaviors (FUEL) trial: Protocol for a cohort study harnessing digital health tools to phenotype dietary non-adherence behaviors during lifestyle intervention. Digit Health. 2024 Aug 21;10:20552076241271783. doi: 10.1177/20552076241271783. eCollection 2024 Jan-Dec. PMID 39175923